CLINICAL TRIAL: NCT06623955
Title: A Comparative Study of Maternal Serum Stathmin-1 Levels in Pregnancies With Preeclampsia, Severe Preeclampsia, and Healthy Controls
Brief Title: Maternal Serum Stathmin-1 Levels in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Bolluk, MD, Başakşehir Çam & Sakura City Hospital
Other Study IDs: Stathmin-1Study
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Control): This group consists of pregnant women who do not have pre-eclampsia or severe pre-eclampsia. These participants will be matched to the case group based on relevant characteristics such as age, gestational age, and other demographic factors.
- Group 2 (Case - Pre-eclampsia): This group consists of pregnant women diagnosed with pre-eclampsia and severe preeclampsia.

SUMMARY:
This study investigates maternal serum Stathmin-1 (STMN-1) levels in pregnancies complicated by preeclampsia and severe preeclampsia, compared to healthy pregnancies. The aim is to explore potential differences in STMN-1 levels among these groups to better understand its role in preeclampsia pathophysiology. Maternal serum STMN-1 levels will be measured between 32-34 weeks of gestation, and patients will be monitored until delivery to assess whether they develop preeclampsia or severe preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Preeclampsia: Defined by New-onset hypertension (Systolic Blood Pressure ≥140 mmHg and/or Diastolic Blood Pressure ≥90 mmHg) after 20 weeks of gestation, with or without proteinuria.
* Clinical diagnosis of Severe Preeclampsia: Defined by criteria such as severe hypertension (systolic BP ≥160 mmHg or diastolic BP ≥110 mmHg), organ dysfunction (renal insufficiency, liver involvement, neurological complications), thrombocytopenia, pulmonary edema, or fetal growth restriction.
* Control Group: Healthy pregnancies without preeclampsia

Exclusion Criteria:

* Multiple Pregnancies
* Pregestational Diabetes
* Chronic Hypertension
* Systemic Diseases (Chronic kidney disease, autoimmune diseases)
* Fetal Anomalies
* Premature Rupture of Membranes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The groups in this study will be selected consists of pregnant women receiving care at a referral center for maternal care.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Maternal Serum Stathmin-1 | Up to 8 weeks (Patients will be followed from inclusion in the study until the end of their pregnancy.)
  To compare Stathmin-1 Levels between the pre-eclampsia and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)